CLINICAL TRIAL: NCT03223857
Title: Visual Performance of Multifocal Intraocular Lenses Following Removal of the Crystalline Lens
Brief Title: To Evaluate the Visual Performance After Bilateral Implantation of Multifocal Intraocular Lenses
Status: Completed | Type: Observational
Sponsor: University Clinic Frankfurt (Other)
Responsible Party: Principal Investigator, Myriam Böhm, MD, Professor Dr. med. Thomas Kohnen, University Clinic Frankfurt
Other Study IDs: 102/13
Record Dates: First submitted 2017-07-18; First posted 2017-07-21 (Actual); Last update posted 2019-03-25 (Actual); Status verified 2019-03

CONDITIONS: Visual Acuity
Keywords: visual outcomes; multifocal intraocular lens; patient satisfaction; spectacle independence
MeSH Terms: conditions — Patient Satisfaction

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 3 Months
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Procedure: Femtosecond-laser-assisted lens exchange — Bilateral implantation of multifocal intraocular lens (MIOL) following femtosecond-laser-assisted lens exchange

SUMMARY:
To evaluate the visual performance after bilateral implantation of multifocal intraocular lenses.

DETAILED DESCRIPTION:
This study evaluates the visual performance after bilateral implantation of multifocal intraocular lenses (IOL). This prospective study is performed at the department of Ophthalmology, Goethe University, Frankfurt, Germany.

Patients who received bilateral implantation of a multifocal intraocular lens pre-enrollment were included consecutively. Exclusion criteria were previous ocular surgeries excluding cataract surgery and refractive lens exchange, regular corneal astigmatism of >1.5 diopter, and ocular pathologies or corneal abnormalities. At 3 months postoperative examination included manifest refraction; monocular and binocular uncorrected (UCVA) and distance-corrected (DCVA) visual acuity in at far, intermediate at near distance (logMAR); slit-lamp examination. 3 months postoperatively defocus testing, binocular contrast sensitivity (CS) under photopic and mesopic conditions, and a questionnaire on subjective quality of vision, optical phenomena, and spectacle independence were performed.

ELIGIBILITY:
Inclusion Criteria:

* bilateral cataract surgery or refractive lens exchange with the implantation a multifocal intraocular lens
* a regular corneal astigmatism < 1.5 D measured with Pentacam (Oculus, Wetzlar, Germany)

Exclusion Criteria:

* other previous ocular surgeries
* ocular pathologies
* corneal abnormalities
* endothelial cell count below 2000/mm²

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Patients who received bilateral cataract surgery or refractive lens exchange with the implantation of a multifocal intraocular lens
Sampling Method: Non-Probability Sample
Enrollment: 60 (Actual)
Dates: Start 2013-04-09 (Actual); Primary Completion 2018-12-23 (Actual); Study Completion 2019-03-23 (Actual)

PRIMARY OUTCOMES:
Best corrected visual acuity at intermediate distance | Measured 3 month after lens surgery
  Monocular and binocular corrected visual acuity at intermediate distance measured in logMAR 3 month after lens surgery

SECONDARY OUTCOMES:
Best corrected visual acuity at far distance | Measured 3 month after lens surgery
  Monocular and binocular best corrected visual acuity at far distance measured in logMAR 3 month after lens surgery
Best corrected visual acuity at near distance | Measured 3 month after lens surgery
  Monocular and binocular best corrected visual acuity at near distance measured in logMAR 3 month after lens surgery
Uncorrected visual acuity at far distance | Measured 3 month after lens surgery
  Monocular and binocular uncorrected visual acuity at far distance measured in logMAR 3 month after lens surgery
Uncorrected visual acuity at intermediate distance | Measured 3 month after lens surgery
  Monocular and binocular uncorrected visual acuity at intermediate distance measured in logMAR 3 month after lens surgery
Uncorrected visual acuity at near distance | Measured 3 month after lens surgery
  Monocular and binocular uncorrected visual acuity at near distance measured in logMAR 3 month after lens surgery
Binocular contrast sensitivity (CS) under photopic, mesopic, and mesopic with glare lighting conditions | Measured 3 month after lens surgery
  Binocular contrast sensitivity (CS) was measured under photopic, mesopic (0.167 cd/m²), and mesopic with glare lighting conditions by means of the "Frankfurt-Freiburg Contrast and Acuity Test System" (FF-CATS)
Defocus curve testing | Measured 3 month after lens surgery
  Defocus curve (monocular and binocular) was tested from -5.0 D to +2.0 D in 0.5 D steps under photopic lighting conditions (ETDRS).

CONTACTS AND LOCATIONS:
Overall Officials: Thomas Kohnen, Professor, Study Chair — Goethe University Clinic Frankfurt
Locations (1):
- Department of ophthalmology University clinic Frankfurt, Frankfurt am Main, Hesse, Germany

IPD SHARING:
Plan to Share IPD: No